CLINICAL TRIAL: NCT06665295
Title: Randomized Controlled Trial of a Supportive Care Digital Application (THRIVE-CAR-T) for Patients Receiving CAR-T Cell Therapy
Brief Title: THRIVE-CAR-T Digital App
Acronym: THRIVE-CAR-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick C. Johnson, MD (Other)
Responsible Party: Sponsor-Investigator, Patrick C. Johnson, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-428
Record Dates: First submitted 2024-10-24; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: CAR T-Cell Therapy
Keywords: car-t cell therapy; digital application; mobile application; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Usual care at our institution involves a teaching visit with a nurse navigator and written handouts.
- THRIVE-CAR-T plus usual care (Experimental): Patients receiving the THRIVE-CAR-T intervention will receive usual care and will use the THRIVE-CAR-T digital application on an iPad when planned to receive CAR-T.
  Interventions: Behavioral: THRIVE-CAR-T

INTERVENTIONS:
Behavioral: THRIVE-CAR-T — The intervention will begin several weeks prior to CAR-T cell therapy and will continue up until 30 days post CAR-T cell therapy. THRIVE-CAR-T is an educational and interactive digital application on an iPad for patients as they navigate receiving CAR-T. THRIVE-CAR-T is self-administered and provides education about the CAR-T cell therapy process, with several features to promote coping skills training informed by various well-established supportive psychotherapy strategies (e.g., cognitive behavior therapy, mindfulness, positive psychology), engagement, and health behavior change including gamification strategies, videos of patients who received CAR-T, and optional content.
  Arms: THRIVE-CAR-T plus usual care

SUMMARY:
The goal of this clinical trial is to learn if a digital mobile application called THRIVE-CAR-T is helpful for the care of patients undergoing CAR-T cell therapy. The main question[s] it aims to answer are whether the THRIVE-CAR-T app is feasible and acceptable to patients.

DETAILED DESCRIPTION:
This pilot randomized controlled trial aims to examine the feasibility, acceptability, and preliminary effects of a supportive care digital app (THRIVE-CAR-T) versus usual care in patients receiving chimeric antigen receptor T-cell therapy (CAR-T). The primary objective of the study is to determine if THRIVE-CAR-T is feasible and acceptable to patients. The exploratory objective is to assess the preliminary effects of THRIVE-CAR-T for improving patient-reported quality of life (QOL), psychological distress, and self efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Ability to understand English
3. Diagnosis of a hematologic malignancy
4. Receiving autologous CAR-T at MGH with an FDA approved cellular therapy product

Exclusion Criteria:

1. Impaired cognition or uncontrolled mental illness that prohibits the ability to provide informed consent based on the oncology clinician assessment
2. Already participating in another supportive care clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Through study completion, an average of 2 years
  Feasibility is defined based on the rate of patient enrollment. THRIVE-CAR-T will be deemed feasible if rates of enrollment are >= 60%, and among those enrolled and randomized to THRIVE-CAR-T, 60% complete 3 out of 5 modules. For patients who either die prior to the end of the intervention or are admitted to the intensive care unit (ICU), the latter definition of feasibility will be completion of 60% of expected modules at the time of clinical deterioration.

SECONDARY OUTCOMES:
Acceptability | Through study completion, an average of 2 years
  THRIVE-CAR-T will be deemed acceptable if at least 80% of patients report THRIVE-CAR-T is acceptable based upon a rating of "Somewhat comfortable" or "Very comfortable" on a 4 point Likert scale single question when asked about whether they feel comfortable with the intervention.
Quality of life | From enrollment until 90 days after CAR-T cell therapy
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy-General (FACT-G). The FACT-G is a 27-item measure consisting of four subscales assessing well-being across four domains (physical, functional, emotional, and social) during the preceding week. Scores range from 0 to 108, with higher scores indicating better QOL
Anxiety symptoms | From enrollment until 90 days after CAR-T cell therapy
  Anxiety symptoms will be assessed using the Hospital Anxiety and Depression Scale (HADS), a 14-item measure with two separate subscales to evaluate symptoms of anxiety and depression. Scores on each subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety or depression.
Depression symptoms | From enrollment until 90 days after CAR-T cell therapy
  Depression symptoms will be assessed using the Hospital Anxiety and Depression Scale (HADS), a 14-item measure with two separate subscales to evaluate symptoms of anxiety and depression. Scores on each subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety or depression
PTSD symptoms | From enrollment until 90 days after CAR-T cell therapy
  PTSD symptoms will be assessed using the Post-traumatic Stress Disorder Checklist-Civilian Version, a17-item PTSD Checklist that evaluates the severity of PTSD symptoms. Scores range from 0-68. Higher scores on the PCL indicate worse PTSD symptoms, with a cutoff of 32 or greater denoting clinically significant PTSD symptoms

OTHER OUTCOMES:
Self-efficacy | From enrollment until 90 days after CAR-T cell therapy
  Self-efficacy will be assessed using the Cancer Self-efficacy Scale (CASE), a commonly utilized measure to assess patients' confidence in managing the impact of their illness. Scores range from 12-48, with higher scores denoting better self-efficacy.
Coping | From enrollment until 90 days after CAR-T cell therapy
  Coping will be assessed using the Measure of Current Status Part A (MOCS-A), a 13-item measure to assess the self-perceived status on several coping skills such as relaxation, cognitive restructuring, and assertive communication. Scores range from 0-52, wither scores denoting greater coping ability.
Knowledge about CAR-T cell therapy | From enrollment until 90 days after CAR-T cell therapy
  Knowledge will be assessed with a Knowledge assessment, where patients will complete nine true/false questions and one multiple choice question to assess patients' knowledge regarding CAR T-cell therapy, with each question worth 1 point for a possible total of 10 points, as done in prior work. Scores range from 0-10, with higher scores denoting greater knowledge.
Usability of THRIVE-CAR-T | From enrollment until 30 days after CAR-T cell therapy
  Usability of THRIVE-CAR-T will only be assessed in those randomized to THRIVE-CAR-T). We will use the system usability scale at day 30 to assess the usability of THRIVE-CAR-T. Scores range from 0-100, with higher scores denoting greater usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be made available upon email request to the principal investigator.